CLINICAL TRIAL: NCT03867227
Title: Non-pharmacological Prevention of Stroke in Patients With Non-valvular Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Collaborators: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government); National Research Center of Surgery, Russia (Other Government); I.M. Sechenov First Moscow State Medical University (Other); Medical and Rehabilitation center (Unknown)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 2018/10/21
Record Dates: First submitted 2019-02-06; First posted 2019-03-07 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
Keywords: left atrial appendage; LAA occluder; thromboembolic prophylaxis; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: left atrial appendage occluder implantation — all patients will get implantation of LAA occluder

SUMMARY:
Left atrial appendage (LAA) occlude devices are used for over ten years. According to current data efficiency and safety of this approach at least comparable with pharmacological prevention of stroke in patients with non-valvular atrial fibrillation.

However, to date, LAA occluder implantation is not recommended as an alternative for conservative therapy and reserved for patients with contraindications for oral anticoagulants only. In the same time, long-term follow-up of patients enrolled in clinical trials and data from registries showed that LAA occlude device implantation as an alternative to oral anticoagulation could reduce drug load, decrease complexity and cost of treatment and thus improve patients' quality of life, and potentially may reduce the risk of death. The aim of our study is to investigate the risk of all-cause death, stroke, and bleedings in patients with LAA occluder implanted as an alternative to anticoagulant therapy.

Three hundred patients with atrial fibrillation will undergo LAA occluder implantation. For LAA occluder sizing transesophageal echocardiography (TEE), CT and LAA angiography will be performed. The follow-up period will be 36 months. The incidence of all-cause death, stroke, bleeding BARC≥2, device-related complications and QOL will be investigated.

The patients will be followed in the clinic at three and six months, and then at 12, 24 and 36 months, the telephone calls for getting information about endpoints events will be done. Additional in clinic visits will be scheduled if the late complications will be suspected.

TEE will be performed at three and six months to check for device leak, displacement and thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with paroxysmal/persistent/permanent atrial fibrillation
* CHA2DS2VASc score ≥2 for male and ≥3 for female
* Without contraindications to anticoagulation therapy

Exclusion Criteria:

* LAA thrombosis
* mechanical prosthetic heart valve
* moderate or severe mitral valve stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years old with atrial fibrillation and high risk for tromboembolic events
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with Composite of death, stroke, clinically significant bleeding event (>_2 class according to BARC criteria), device leak, device displacement or device thrombosis with the first event for a given patient is taken into account | 36 months
  a clinically significant bleeding event is >_2 class according to Bleeding Academic Research Consortium (BARC) criteria bleeding

SECONDARY OUTCOMES:
device thrombosis during first 6 months | 6 months
  device thrombosis detected by transesophageal echocardiography during first 6 months of follow-up
device dislocation | 36 months
  number of patients who would have device dislocation
any bleed | 36 months
  total number of patients who would have any bleeding event
bleeding BARC ≥2 | 36 months
  total number of patients who would have bleeding event with the grade BARC ≥2
device leak and displacement during first 6 months | 6 months
  device leak detected by transesophageal echocardiography during first 6 months after implantation or device displacement during the same time period
any adverse events during 7 days after LAA occluder implantation | 7 days
  any adverse events related to the device implantation during the first 7 days after implantation
change in QOL SF 36 between baseline and final visit | Assessed at baseline and 6-month follow-up visits
  change in quality of life (QOL) by Short Form (SF) 36 Health Survey between baseline and follow-up visits
  SF 36 is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health. 0-100 scale are using to access each domain. lower the score the more disability.
the percent of patients in whom long -term anticoagulation therapy would add during follow-up | 36 months
  number of patients who would require adding permanent anticoagulant therapy for any reason during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Karapet Davtyan, Principal Investigator — National Research Center for Preventive Medicine
Locations (1):
- . National Research Center for Preventive Medicine of the Ministry of Health, Moscow, Russia